CLINICAL TRIAL: NCT03369639
Title: Observational Study of Dronabinol Treatment for Depression and/or Anxiety in Older Patients
Brief Title: Study of Dronabinol Treatment for Depression and/or Anxiety in Older Patients
Status: Withdrawn | Type: Observational
Why Stopped: Due to prohibitively high drug cost, physicians were not prescribing the drug.
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Brent Forester, Director, Geriatric Psychiatry Research Program and Geriatric Mood Disorders Research Program, Mclean Hospital
Other Study IDs: 2017P001930
Record Dates: First submitted 2017-11-14; First posted 2017-12-12 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Depression, Anxiety
Keywords: late life; THC; depression; anxiety; dronabinol
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational study evaluating the safety and efficacy of dronabinol for the treatment of anxiety and/or depression in older adults. Participants who are prescribed dronabinol as part of a voluntary inpatient stay in McLean's Division of Geriatric Psychiatry will be interviewed about their mood and cognition on a weekly basis while on dronabinol.

DETAILED DESCRIPTION:
Recently there has been renewed interest in potential alternative medical applications of cannabis/THC and medical marijuana is now legalized in 23 states and the District of Columbia. Acute effects of THC can include subjective feelings of euphoria, relaxation, and sedation, and clinicians noted that THC is well tolerated for its approved indications. Given these subjective effects and relatively benign safety profile, some physicians have used dronabinol (synthetic THC) "off-label" to treat depression and/or anxiety.

The investigators are doing this research to better understand how effective dronabinol treatment is when prescribed for depression and/or anxiety in older patients. The investigators also want to find out if dronabinol is safe to take without causing too many side effects. Dronabinol is is approved by the U.S. Food and Drug Administration (FDA) to treat loss of appetite in chemotherapy patients, but dronabinol is not approved by the FDA to treat depression and/or anxiety. Through research questionnaires on mood and cognition, the investigators can gather information that will help demonstrate how effective dronabinol treatment is at treating depression and/or anxiety.

ELIGIBILITY:
Inclusion Criteria:

1. 50-89 years old (inclusive)
2. Inpatient on the Older Adult Unit in South Belknap 1 at McLean Hospital
3. Initiating dronabinol therapy for the treatment of any Diagnostic and Statistical Manual (DSM) 5 Major Depression or Anxiety Disorder Diagnosis
4. Ability to provide informed consent
5. Must be fluent in English

Exclusion Criteria:

1. Delirium as determined by the Confusion Assessment Method (CAM)
2. Serious or unstable medical illness, including cardiovascular, hepatic, renal, respiratory, endocrine, neurologic or hematologic disease, which might confound assessment of safety outcomes
3. Seizure disorder
4. Diagnosis of bipolar depression, Major depression with psychotic features, schizophrenia, schizoaffective disorder, dementia
5. Use of dronabinol or marijuana in the last year
6. Prescription of lithium or anticonvulsant medications (except gabapentin)
7. Patient currently admitted involuntarily to McLean Hospital

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the Mood Disorder inpatient unit within the Division of Geriatric Psychiatry at McLean Hospital. These older patients will have a diagnosis of major depression and/or anxiety and have agreed to begin dronabinol treatment after recommendation by the attending physician.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Efficacy against depression as measured by the MADRS | Weekly, from baseline prior to first dose for 2 weeks
  Assessed via the Montgomery Asberg Depression Rating Scale (MADRS). The MADRS score ranges from 0 (least depressed) to 60 (most depressed).
Efficacy against anxiety as measured by the HAM-A | Weekly, from baseline prior to first dose for 2 weeks
  Assessed via the Hamilton Anxiety Rating Scale (HAM-A). The HAM-A score ranges from 0 (no present anxiety) to 56 (maximum anxiety score).

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse effects (Safety) | Weekly, from baseline prior to first dose for 2 weeks
  Assessed by tracking and recording of adverse events and serious adverse events, and interviews about drug effects
Cognition | At baseline prior to first dose and at 2 weeks
  Assessed by administration of the Montreal Cognitive Assessment (MoCA) at baseline and after 2 weeks of dronabinol. MoCA score ranges from 0 (most cognitively impaired) to 30 (least impaired).
Efficacy against depression as measured by the GDS | Weekly, from baseline prior to first dose for 2 weeks
  Assessed by administration of the Geriatric Depression Scale (GDS). The GDS score ranges from 0 (least depressed) to 15 (most depressed).
Efficacy against anxiety as measured by the GAD-7 | Weekly, from baseline prior to first dose for 2 weeks
  Assessed by administration of the Generalized Anxiety Disorder--7 (GAD-7) scale. The GAD-7 score ranges from 0 (no anxiety) to 21 (highest, severe anxiety).

CONTACTS AND LOCATIONS:
Overall Officials: Brent P Forester, MD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States